CLINICAL TRIAL: NCT06600893
Title: A Single-Blind, Sham-Controlled, Randomized, Prospective Study Characterizing Erectile Tissue Ultrasound Changes Resulting From Low Intensity Penile Shockwave Treatment With Urogold 100™
Brief Title: Sham-Controlled Prospective Study Characterizing Erectile Tissue Ultrasound Changes Resulting From Penile LiSWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego Sexual Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SDSM-2019-02.1
Record Dates: First submitted 2024-09-14; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Erectile Dysfunctions
Keywords: low intensity shockwave therapy; erectile dysfunction; grayscale ultrasound; duplex Doppler ultrasound; erectile tissue homogeneity/inhomogeneity
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: Sham group crosses over to active treatment while active group does a second follow up assessment without additional treatment intervention
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant is placed behind a screen wearing headphones so they cannot see if the noise of shocking is coming from the shockwave device or from the recording playing on a bluetooth speaker as applicator is placed on the various locations for treatment with energy or simulated sham treatment without energy. Outcomes are assessed without identification of whether the assessment is after active or sham treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Sham Arm 1-Simulated Low Intensity Shockwave Therapy (Sham Comparator): Using the shockwave device, 5000 simulated low intensity shockwave therapy delivered week 0, week 3, week 6
  Interventions: Device: Sham
- Active Arm 1- Low Intensity Shockwave Therapy (Experimental): Using the shockwave device, 5000 low intensity shockwave therapy delivered week 0, week 3, week 6
  Interventions: Device: Low intensity shockwave therapy (LiSWT)
- Sham Arm 2 - Simulated Low Intensity Shockwave Therapy (Sham Comparator): Using the shockwave device, 5000 simulated low intensity shockwave therapy delivered week 0, 3000 week 1, 3000 week 3, 5000 week 6, 3000 week 7, 3000 week 8
  Interventions: Device: Sham
- Active Arm 2 - Low Intensity Shockwave Therapy (Experimental): Using the shockwave device, 5000 low intensity shockwave therapy delivered week 0, 3000 week 1, 3000 week 3, 5000 week 6, 3000 week 7, 3000 week 8
  Interventions: Device: Low intensity shockwave therapy (LiSWT)

INTERVENTIONS:
Device: Low intensity shockwave therapy (LiSWT) — The Urogold100™ uses electrohydraulic technology to generate low intensity shockwave energies in ranges of 0.1 - 0.18 mJ/mm2 (using 0.9 - 0.12 mJ/mm2 in this study) associated with biologic activities of stimulation of mechanosensors, activation of neo-angiogenesis processes, recruitment and activation of stem cell progenitor cells, improvement of microcirculation, nerve regeneration, remodeling of erectile tissue with increase in the muscle/collagen ratio and reducing inflammatory and cellular stress responses. The device uses the parabolic applicator OP 155 that generates a plasma-driven detonation resulting in a shockwave with a broad and widely-stretched 5 megapascal therapeutic volume. Due to the absence of a concentrated focus, a 14 mm wide shockwave is delivered to the erectile tissue with up to 30 mm penetration. LiSWT is delivered to Active Arms 1 and 2 per protocol. After unblinding at the first follow up visit, participants in Sham Arms 1 and 2 receive active LiSWT treatment
  Other Names: SoftWave TRT/UroGold 100MTS; Parabolic applicator OP 155
  Arms: Active Arm 1- Low Intensity Shockwave Therapy; Active Arm 2 - Low Intensity Shockwave Therapy
Device: Sham — With the Urogold 100 turned on and with the participant wearing headphones and blinded by a pulled curtain the applicator is applied in a similar manner to when it is active treatment and the sound of shockwave playing in a blue tooth speaker the participant believes he is receiving active treatment but zero energy is delivered.
  Arms: Sham Arm 1-Simulated Low Intensity Shockwave Therapy; Sham Arm 2 - Simulated Low Intensity Shockwave Therapy

SUMMARY:
The primary goal of this single blind, prospective sham-controlled clinical trial is to assess safety and efficacy of low intensity shockwave therapy (LiSWT) to improve erectile function in men 21-80 years of age with erectile dysfunction naive to radial ballistic acoustic wave and LiSWT. The main questions it aims to answer are:

* Does homogeneity/inhomogeneity of corporal cavernosal tissue improve using Grayscale ultrasound (GUS) when comparing sham to active treatment groups?
* Do peak systolic velocity (PSV) and end diastolic velocity (EDV) improve using color duplex Doppler ultrasound when comparing sham to active treatment groups?
* Do the International Index of Erectile Function (IIEF), its erectile function domain (IIEF-EF) and question 3 of the Sexual Encounter Profile (SEP) improve comparing sham to active treatment groups?

DETAILED DESCRIPTION:
This is a single site sham-controlled clinical trial to be conducted at San Diego Sexual Medicine in San Diego, California. Subjects meeting inclusion and exclusion criteria will be randomized to one of two arms, each 2:1 active to sham, treated in 3-week cycles. Arm 1 consists of 5000 shocks the first week and two weeks off for each of three treatment cycles. Arm 2 is made up of 5000 shocks the first week and 3000 active shocks the second and third weeks followed by three weeks without treatment, and then 5000, 3000 and 3000 shocks again over the next three weeks. Each of these is followed by the first follow-up visit at 20 weeks after the first treatment, when GUS and DUS is repeated and validated instruments completed, at which time treatment will be unblinded. SEP diaries will be completed during sexual activity in the screening period and during the 4 weeks prior to the follow up visit. Those subjects assigned to sham will be crossed over to the opposite arm for active treatment (arm 1 sham goes to arm 2 open label and arm 2 sham to arm 1 open label) and begin active treatment with decreased intervals between shocks and therefore decreased number of shocks needed, with 3500 rather than 5000 shocks and 2000 rather than 3000 shocks at a lower frequency at that visit after completing the follow up procedures. Subjects assigned initially to the active arm will have a second follow up 32 weeks after the first treatment, and complete SEP diaries during the 4 weeks preceding this visit. GUS and DUS is performed and validated instruments completed at the last follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Subject provides written informed consent and HIPAA authorization before any study procedures are conducted;
2. Subject is male;
3. Subject is aged 21-80 years;
4. Subject is in a relationship with a female partner for at least 3 months;
5. Subject has a body mass index (BMI) < 37 kg/m2;
6. Subject has erectile dysfunction;
7. Subject has testosterone ≥ 300;
8. Subject has a prostate specific antigen (PSA) < 4.0;
9. Subject is willing to attempt sexual activity at least 4 times during the screening period and 4 weeks before each follow-up visit;
10. Subject is willing to stop all erectile function aids (e.g. prescription and non-prescription medications, injections, vacuum erection devices, constriction ring) during the screening period and 4 weeks before each follow-up visit;
11. Subject agrees to comply with the study procedures and visits.

Exclusion Criteria:

1. Subject has been treated with acoustic wave previously;
2. Subject has a pacemaker or implanted defibrillator;
3. Subject has clinically significant findings on physical examination;
4. Subject has sciatica or severe back pain;
5. Subject has uncontrolled hypertension;
6. Subject has uncontrolled hypogonadism;
7. Subject is unwilling to maintain testosterone replacement therapy if currently using testosterone to treat hypogonadism;
8. Subject scores ≥ 26 on the IIEF;
9. Subject has homogenous corpora cavernosa on grey scale ultrasound;
10. Subject has any chronic medical condition or psychologic disorder that the Principal Investigator feels makes him ineligible for the study;
11. Subject has lesions or active infections on the penis or perineum;
12. Subject is unwilling to remove piercings from the genital region;
13. Subject has a history of substance abuse within 12 months prior, or consuming > 14 alcoholic drinks per week;
14. Subject has received an investigational drug within 30 days prior to signing consent;
15. Subject has received platelet rich plasma (PRP) within 3 months of signing consent;
16. Subject has received stem cell within 6 months of signing consent;
17. Subject has any condition or exhibits behavior that indicates to the Principal Investigator that the Subject is unlikely to be compliant with study procedures and visits.

Ages: 21 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants had to be anatomically a male and identity as a male.
Enrollment: 35 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2023-04-07 (Actual)

PRIMARY OUTCOMES:
Grayscale ultrasound (GUS) | Baseline to follow up visit 1 at week 20, and follow up visit 2 at week 32 for those assigned initially to the active arm and week 40 to those initially assigned to sham
  Changes from low intensity shockwave treatment using Grayscale ultrasound to assess erectile tissue homogeneity of the corpora cavernosa comparing sham and active treatment groups
Duplex Doppler ultrasound (DUS) | Baseline to follow up visit 1 at week 20, and follow up visit 2 at week 32 for those assigned initially to the active arm and week 40 to those initially assigned to sham
  Changes from low intensity shockwave treatment in peak systolic velocity (PSV) and end diastolic velocity (EDV) using color duplex Doppler ultrasound comparing sham and active treatment groups

SECONDARY OUTCOMES:
International Index of Erectile Function (IIEF) | Baseline to follow up visit 1 at week 20, and follow up visit 2 at week 32 for those assigned initially to the active arm and week 40 to those initially assigned to sham
  Changes in IIEF, a validated patient reported outcome instrument used to assess sexual function will be compared from baseline to both follow up visit. This has a 4 week recall.
IIEF Erectile Function Domain (IIEF-EF) | Baseline to follow up visit 1 at week 20, and follow up visit 2 at week 32 for those assigned initially to the active arm and week 40 to those initially assigned to sham
  Changes in the erectile function domain, IIEF-EF, used specifically to assess erectile function, will be compared from baseline to both follow up visit. This is a 4 week recall.
Sexual Encounter Profile (SEP) | Completed over the 4 week screening period, and during the 4 weeks prior to each follow up
  The SEP diary is a standard assessment completed by a participant after each attempt at sexual activity.

OTHER OUTCOMES:
International Prostate Symptom Score (IPSS) | Baseline to follow up visit 1 at week 20, and follow up visit 2 at week 32 for those assigned initially to the active arm and week 40 to those initially assigned to sham
  The IPSS is a validated patient reported outcome instrument to assesses lower urinary tract symptoms, comparing baseline to follow up visits in active and sham groups.

CONTACTS AND LOCATIONS:
Overall Officials: Irwin Goldstein, MD, Principal Investigator — San Diego Sexual Medicine
Locations (1):
- San Diego Sexual Medicine, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
The research is from a small medical practice without the manpower, financial or technical support from a larger institution or industry to enter data into a data repository.

REFERENCES:
- [Background] Kitrey ND, Vardi Y, Appel B, Shechter A, Massarwi O, Abu-Ghanem Y, Gruenwald I. Low Intensity Shock Wave Treatment for Erectile Dysfunction-How Long Does the Effect Last? J Urol. 2018 Jul;200(1):167-170. doi: 10.1016/j.juro.2018.02.070. Epub 2018 Mar 1. PMID 29477719
- [Background] Kalyvianakis D, Hatzichristou D. Low-Intensity Shockwave Therapy Improves Hemodynamic Parameters in Patients With Vasculogenic Erectile Dysfunction: A Triplex Ultrasonography-Based Sham-Controlled Trial. J Sex Med. 2017 Jul;14(7):891-897. doi: 10.1016/j.jsxm.2017.05.012. PMID 28673433
- [Background] Kalyvianakis D, Memmos E, Mykoniatis I, Kapoteli P, Memmos D, Hatzichristou D. Low-Intensity Shockwave Therapy for Erectile Dysfunction: A Randomized Clinical Trial Comparing 2 Treatment Protocols and the Impact of Repeating Treatment. J Sex Med. 2018 Mar;15(3):334-345. doi: 10.1016/j.jsxm.2018.01.003. Epub 2018 Feb 1. PMID 29396020
- [Background] Sokolakis I, Hatzichristodoulou G. Clinical studies on low intensity extracorporeal shockwave therapy for erectile dysfunction: a systematic review and meta-analysis of randomised controlled trials. Int J Impot Res. 2019 May;31(3):177-194. doi: 10.1038/s41443-019-0117-z. Epub 2019 Jan 21. PMID 30664671
- [Background] Sokolakis I, Dimitriadis F, Teo P, Hatzichristodoulou G, Hatzichristou D, Giuliano F. The Basic Science Behind Low-Intensity Extracorporeal Shockwave Therapy for Erectile Dysfunction: A Systematic Scoping Review of Pre-Clinical Studies. J Sex Med. 2019 Feb;16(2):168-194. doi: 10.1016/j.jsxm.2018.12.016. PMID 30770067
- [Background] Rizk PJ, Krieger JR, Kohn TP, Pastuszak AW. Low-Intensity Shockwave Therapy for Erectile Dysfunction. Sex Med Rev. 2018 Oct;6(4):624-630. doi: 10.1016/j.sxmr.2018.01.002. Epub 2018 Mar 22. PMID 29576441
- [Background] Ruffo A, Capece M, Prezioso D, Romeo G, Illiano E, Romis L, Di Lauro G, Iacono F. Safety and efficacy of low intensity shockwave (LISW) treatment in patients with erectile dysfunction. Int Braz J Urol. 2015 Sep-Oct;41(5):967-74. doi: 10.1590/S1677-5538.IBJU.2014.0386. PMID 26689523
- [Derived] Goldstein SW, Kim NN, Goldstein I. Randomized trial of low intensity shockwave therapy for erectile dysfunction utilizing grayscale ultrasound for analysis of erectile tissue homogeneity/inhomogeneity. Transl Androl Urol. 2024 Oct 31;13(10):2246-2267. doi: 10.21037/tau-24-338. Epub 2024 Oct 28. PMID 39507857